CLINICAL TRIAL: NCT00891826
Title: Omega-3 Fatty Acids in Bipolar Patients With a Low Omega-3 Index and Reduced Heart Rate Variability: the "BIPO-3" Trial
Brief Title: Omega-3 Fatty Acids in Bipolar Patients With a Low Omega-3 Index and Reduced Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, W. Emanuel Severus, M.D., University Hospital Dresden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPAX 103
Record Dates: First submitted 2009-04-28; First posted 2009-05-01 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Bipolar Disorders
Keywords: Bipolar disorders; Omega-3 fatty acids; Heart rate
MeSH Terms: conditions — Bipolar Disorder | interventions — Fatty Acids, Omega-3; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corn oil (Placebo Comparator)
  Interventions: Dietary Supplement: Corn oil
- Omega-3 fatty acids (Experimental)
  Interventions: Dietary Supplement: Omega-3 fatty acids (EPAX 6015 TG)

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids (EPAX 6015 TG) — The study drug is a food supplement called EPAX 6015 TG. One capsule of EPAX 6015 TG contains 530 mg of EPA (eicosapentaenoic acid) and 150 mg of DHA (docosahexaenoic acid), provided as triglycerides. For the entire study period (12 weeks) patients will receive 4 capsules of EPAX 6015 TG per day.
  Arms: Omega-3 fatty acids
Dietary Supplement: Corn oil — The corn oil capsules look exactly the same as the capsules containing omega-3 fatty acids. For the entire study period patients will receive 4 capsules of corn oil per day.
  Arms: Corn oil

SUMMARY:
This study sets out to test the hypothesis that parameters of heart rate variability, as a non-invasive measure of cardiovascular risk, can be improved by the addition of omega-3 fatty acids in euthymic bipolar patients with a low omega-3 index and reduced heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet the DSM-IV criteria for bipolar disorders, in remission
2. Age: 18 - 65 years
3. Low omega-3 index (<5%)
4. SDNN < 60 msec
5. Subjects must have adequate fluency in German or English to complete baseline and follow-up interviews and fill out the Beck Depression Inventory
6. Stable psychotropic medication for at least 2 weeks
7. Subjects must be able to give written informed consent

Exclusion Criteria:

1. Subjects for whom the intake of omega-3 fatty acids is indicated according to recent treatment guidelines
2. Patients on Warfarin
3. Subjects with any acute and life-threatening condition, such as collapse and shock, acute myocardial infarction, stroke, embolism
4. Subjects with significant medical comorbidity
5. Pregnant subjects - due to any possible teratogenic effects of EPAX 6015 TG and corn oil, respectively, on the fetus - and breastfeeding subjects. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded
6. Subjects who, in the investigator's judgement, pose a current significant suicidal or homicidal risk or patients who will not likely be able to comply with the study protocol
7. Subjects fulfilling the DSM-IV diagnostic criteria for current substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
SDNN (msec) | at baseline and after 12 weeks

SECONDARY OUTCOMES:
LF/HF ratio | at baseline and after 12 weeks
Time to new episode | study period (12 weeks)
Mood Rating Scales | at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Severus, M.D., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Department of Psychiatry, University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Berger M, Seemuller F, Voggt A, Obermeier M, Kirchberg F, Low A, Riedel M, von Schacky C, Severus E. Omega-3 fatty acids in bipolar patients with a low omega-3 index and reduced heart rate variability: the "BIPO-3" trial. Int J Bipolar Disord. 2022 Apr 1;10(1):9. doi: 10.1186/s40345-022-00253-9. PMID 35362878